CLINICAL TRIAL: NCT02030600
Title: A Randomised, Double Blind, Cross-over Trial Comparing the Safety and Efficacy of Insulin Degludec and Insulin Glargine, With or Without OADs in Subjects With Type 2 Diabetes (SWITCH 2)
Brief Title: A Trial Comparing the Safety and Efficacy of Insulin Degludec and Insulin Glargine, With or Without OADs in Subjects With Type 2 Diabetes
Acronym: SWITCH 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3998; U1111-1143-7963 (Other: WHO)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD ± OADs followed by IGlar OD ± OADs (Experimental): The trial includes two 32-week treatment periods in a cross-over design. Total trial duration for the individual subjects will be up to 67 weeks.
  Interventions: Drug: insulin degludec; Drug: insulin glargine
- IGlar OD ± OADs followed by IDeg OD ± OADs (Active Comparator): The trial includes two 32-week treatment periods in a cross-over design. Total trial duration for the individual subjects will be up to 67 weeks.
  Interventions: Drug: insulin degludec; Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Administered once daily injected s.c. / subcutaneously (under the skin). Dose is individually adjusted.
Drug: insulin glargine — Administered once daily injected s.c. / subcutaneously (under the skin). Dose is individually adjusted.

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of the trial is to compare the safety and efficacy of insulin degludec (IDeg) and insulin glargine (IGlar) with or without OADs (oral anti-diabetic drugs) excluding SUs (sulfonylureas)/glinides in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Male or female, age at least 18 years at the time of signing informed consent - Subjects fulfilling at least one of the below criteria: a) Experienced at least one severe hypoglycaemic episode within last year (according to the ADA (American Diabetes Association) definition, April 2013), b) Moderate chronic renal failure, defined as glomerular filtration rate 30 - 59 mL/min/1.73 m^2 per CKD-Epi (Chronic Kidney Disease Epidemiology Collaboration) by central laboratory analysis, c) Hypoglycaemic symptom unawareness, d) Exposed to insulin for more than 5 years, e) Recent episode of hypoglycaemia (defined by symptoms of hypoglycaemia and/or episode with low glucose measurement (below or equal to 70 mg/dL [below or equal to 3.9 mmol/L])) within the last 12 weeks prior to Visit 1 (screening) - Type 2 diabetes mellitus (diagnosed clinically) for at least 26 weeks prior to Visit 1 - Current treatment with any basal insulin (OD or BID) ± any combination of OADs (metformin, DPP-4 inhibitor, alpha-glucosidase inhibitor, thiazolidinediones, and SGLT2-inhibitor) for 26 weeks or longer prior to Visit 1 For subjects on BID the total daily dose should be below 75 units - HbA1c (glycosylated haemoglobin) below or equal to 9.5 % by central laboratory analysis - BMI (body mass index) below or equal to 45 kg/m^2 Exclusion Criteria: - Treatment with a bolus insulin separately or contained in an insulin mix product within the last 26 weeks prior to Visit 1 - Use of any other anti-diabetic agent(s) than those stated in the inclusion criteria within the last 26 weeks prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2015-12-04 (Actual); Study Completion 2015-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (135):
- United States (131):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Haleyville, Alabama
  - Novo Nordisk Investigational Site, Montgomery, Alabama
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Costa Mesa, California
  - Novo Nordisk Investigational Site, Downey, California
  - Novo Nordisk Investigational Site, El Cajon, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Hawaiian Gardens, California
  - Novo Nordisk Investigational Site, Huntington Park, California
  - Novo Nordisk Investigational Site, Lincoln, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, North Hollywood, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Pomona, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Rancho Cucamonga, California
  - Novo Nordisk Investigational Site, Rialto, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Tarzana, California
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Newark, Delaware
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Chiefland, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Doral, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Springs, Florida
  - Novo Nordisk Investigational Site, Miramar, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Panama City, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Perry, Georgia
  - Novo Nordisk Investigational Site, Champaign, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, West Des Moines, Iowa
  - Novo Nordisk Investigational Site, Lenexa, Kansas
  - Novo Nordisk Investigational Site, Newton, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Brockton, Massachusetts
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Olive Branch, Mississippi
  - Novo Nordisk Investigational Site, Florissant, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Newington, New Hampshire
  - Novo Nordisk Investigational Site, Morganville, New Jersey
  - Novo Nordisk Investigational Site, Teaneck, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Jackson Heights, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Morganton, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Delaware, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Scottdale, Pennsylvania
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Gaffney, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Pelzer, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Rapid City, South Dakota
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Jackson, Tennessee
  - Novo Nordisk Investigational Site, Johnson City, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Carrollton, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, El Paso, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Humble, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Marshall, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, North Richland Hills, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, Richardson, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sealy, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Victoria, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, Draper, Utah
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Richland, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Martinsburg, West Virginia
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Puerto Rico (4):
  - Novo Nordisk Investigational Site, Carolina
  - Novo Nordisk Investigational Site, Manatí
  - Novo Nordisk Investigational Site, Ponce
  - Novo Nordisk Investigational Site, San Juan

REFERENCES:
- [Background] Chaykin L, Bhargava A, de la Rosa R, Wysham CH, Norgard Troelsen L, Ostoft SH, Philis-Tsimikas A. Effect of Insulin Degludec Versus Insulin Glargine U100 on Hypoglycemia in Hispanic Patients With Type 2 Diabetes: Results From the SWITCH 2 Trial. Clin Diabetes. 2019 Jan;37(1):73-81. doi: 10.2337/cd18-0016. PMID 30705500
- [Result] Wysham C, Bhargava A, Chaykin L, de la Rosa R, Handelsman Y, Troelsen LN, Kvist K, Norwood P. Effect of Insulin Degludec vs Insulin Glargine U100 on Hypoglycemia in Patients With Type 2 Diabetes: The SWITCH 2 Randomized Clinical Trial. JAMA. 2017 Jul 4;318(1):45-56. doi: 10.1001/jama.2017.7117. PMID 28672317
- [Result] Evans M, Mehta R, Gundgaard J, Chubb B. Cost-Effectiveness of Insulin Degludec vs. Insulin Glargine U100 in Type 1 and Type 2 Diabetes Mellitus in a UK Setting. Diabetes Ther. 2018 Oct;9(5):1919-1930. doi: 10.1007/s13300-018-0478-1. Epub 2018 Aug 10. PMID 30097995
- [Result] DeVries JH, Bailey TS, Bhargava A, Gerety G, Gumprecht J, Heller S, Lane W, Wysham CH, Zinman B, Bak BA, Hachmann-Nielsen E, Philis-Tsimikas A. Day-to-day fasting self-monitored blood glucose variability is associated with risk of hypoglycaemia in insulin-treated patients with type 1 and type 2 diabetes: A post hoc analysis of the SWITCH Trials. Diabetes Obes Metab. 2019 Mar;21(3):622-630. doi: 10.1111/dom.13565. Epub 2018 Nov 26. PMID 30362250
- [Result] Heller SR, DeVries JH, Wysham C, Hansen CT, Hansen MV, Frier BM. Lower rates of hypoglycaemia in older individuals with type 2 diabetes using insulin degludec versus insulin glargine U100: Results from SWITCH 2. Diabetes Obes Metab. 2019 Jul;21(7):1634-1641. doi: 10.1111/dom.13708. Epub 2019 Apr 15. PMID 30891886
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 152 sites in the United States.
Groups:
- Insulin Degludec/Insulin Glargine (IDeg/IGlar): Subjects received insulin degludec (IDeg) in treatment period 1 and insulin glargine (IGlar) in treatment period 2. Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IDeg and IGlar were administered in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken at the same time of day throughout the trial. Subjects receiving pre-trial once daily basal insulin were to continue on their pre-trial basal insulin dose. For subjects receiving pre-trial twice daily basal insulin, a 20% reduction of the total daily insulin dose was recommended. Doses of IDeg and IGlar were titrated individually. Adjustment of the dose was performed once weekly based on the mean of 3 preceding daily fasting self-measured plasma glucose (SMPG) values on 3 consecutive days (fasting glycaemic target of 4.0-5.0 mmol/L).
- Insulin Glargine/Insulin Degludec (IGlar/IDeg): Subjects received IGlar in treatment period 1 and IDeg in treatment period 2. Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IGlar and IDeg were administered in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken at the same time of day throughout the trial. Subjects receiving pre-trial once daily basal insulin were to continue on their pre-trial basal insulin dose. For subjects receiving pre-trial twice daily basal insulin, a 20% reduction of the total insulin daily dose was recommended. Doses of IGlar and IDeg were titrated individually. Adjustment of the dose was performed once weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-5.0 mmol/L).
Period: Treatment Period 1
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg)
Started | 361 | 360
Exposed | 356 | 357
Completed | 308 | 315
Not Completed | 53 | 45
Not completed — Adverse Event | 5 | 7
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 11 | 3
Not completed — Protocol Violation | 22 | 17
Not completed — Withdrawal by Subject | 13 | 17
Not completed — Casebook Unsigned | 1 | 0
Not completed — Unclassified | 1 | 0
Period: Treatment Period 2
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg)
Started | 308 | 315
Completed | 283 | 297
Not Completed | 25 | 18
Not completed — Adverse Event | 4 | 4
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 4 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Unclassified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomised subjects. One subject was excluded from the analysis due to unsigned casebook.
Groups:
- Insulin Degludec/Insulin Glargine (IDeg/IGlar): Subjects received IDeg in treatment period 1 and IGlar in treatment period 2. Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IDeg and IGlar were administered in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken at the same time of day throughout the trial. Subjects receiving pre-trial once daily basal insulin were to continue on their pre-trial basal insulin dose. For subjects receiving pre-trial twice daily basal insulin, a 20% reduction of the total daily insulin dose was recommended. Doses of IDeg and IGlar were titrated individually. Adjustment of the dose was performed once weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-5.0 mmol/L).
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg) | Total
Number analyzed (Participants) | 360 | 360 | 720
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.7) | 61.2 (10.3) | 61.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 169 | 338
  Male | 191 | 191 | 382
Glycosylated haemoglobin [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.6 (1.1) | 7.6 (1.1) | 7.6 (1.1)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] — Number of subjects analyzed=355 for IDeg/IGlar arm, 358 for IGlar/IDeg arm and 713 for total.
  mg/dL | 139.2 (53.5) | 134.9 (51.6) | 137.0 (52.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Maintenance Period
Description: Severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe and/or BG confirmed by a plasma glucose value of <56 mg/dL (3.1 mmol/L), with symptoms consistent with hypoglycaemia. Treatment emergent hypoglycaemic episode was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Time Frame: After 16 weeks of treatment, in each treatment period (Week 16-32 and Week 48-64)
Population: The trial followed a cross over design. Descriptive analysis was based on the safety analysis set (subjects receiving at least one dose of the investigational product or its comparator). Number of subjects analysed=subjects with available data for the endpoint as per individual trial products. Statistical analysis was performed on full analysis set
Measure: Number; unit: events
Groups:
- Insulin Degludec (IDeg): Subjects receiving IDeg in treatment period 1 (from treatment sequence IDeg/IGlar) and in treatment period 2 (from treatment sequence IGlar/IDeg). Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IDeg was administered in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken at same time of day throughout the trial. Subjects receiving pre-trial once daily basal insulin were to continue on their pre-trial basal insulin dose. For subjects receiving pre-trial twice daily basal insulin, a 20% reduction of the total daily insulin dose was recommended. Dose of IDeg was titrated individually. Adjustment of dose was performed once weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-5.0 mmol/L).
- Insulin Glargine (IGlar): Subjects receiving IGlar in treatment period 1 (from treatment sequence IGlar/IDeg) and in treatment period 2 (from treatment sequence IDeg/IGlar). Each treatment period consisted of a 16-week titration period and a 16-week maintenance period (total 32 weeks for each treatment period). IGlar was administered in the morning (from waking up to breakfast) or in the evening (from main evening meal to bedtime), as per randomisation and were to be taken at same time of day throughout the trial. Subjects receiving pre-trial once daily basal insulin were to continue on their pre-trial basal insulin dose. For subjects receiving pre-trial twice daily basal insulin, a 20% reduction of the total daily insulin dose was recommended. Dose of IGlar was titrated individually. Adjustment of dose was performed once weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-5.0 mmol/L).
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 632 | 618
events | 353 | 496
Statistical Analysis 1: Comparison: Insulin Degludec (IDeg) vs Insulin Glargine (IGlar); Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 1: Primary analysis: Number of treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the maintenance period; Test type: Superiority or Other; p < 0.0001, Poisson; Treatment ratio = 0.70, 95% CI 2-sided [0.61 to 0.80] — Superiority was considered confirmed if the 95% confidence interval for the rate ratio (IDeg/IGlar) was entirely below 1.0

2. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Nocturnal Hypoglycaemic Episode During the Maintenance Period
Description: Severe or BG confirmed symptomatic nocturnal hypoglycaemic episodes were defined as episodes that were severe and/or BG confirmed by a plasma glucose value of <56 mg/dL (3.1 mmol/L), with symptoms consistent with hypoglycaemia and with time of onset between 00:01 and 05.59 a.m., both inclusive. Treatment emergent hypoglycaemic episode was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Time Frame: After 16 weeks of treatment, in each treatment period (Week 16-32 and Week 48-64)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 632 | 618
events | 105 | 175
Statistical Analysis 1: Comparison: Insulin Degludec (IDeg) vs Insulin Glargine (IGlar); Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 2: Number of treatment-emergent severe or BG confirmed symptomatic nocturnal hypoglycaemic episodes during the maintenance period; Test type: Superiority or Other; p < 0.0001, Poisson; Treatment ratio = 0.58, 95% CI 2-sided [0.46 to 0.74] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Subjects With One or More Severe Hypoglycaemic Episodes During the Maintenance Period
Description: Percentage of subjects who experienced one or more severe hypoglycaemic episodes during the maintenance period. Severe hypoglycaemia (according to the American Diabetes Association 2013 definition): A hypoglycaemic episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose values may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: After 16 weeks of treatment, in each treatment period (Week 16-32 and Week 48-64)
Population: The trial followed a cross over design. Descriptive analysis was based on the safety analysis set. Number of subjects analysed=subjects with available data for the endpoint as per individual trial products. Statistical analysis was performed on subjects in full analysis set with exposure in both maintenance periods.
Measure: Number; unit: percentage of subjects
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 632 | 618
percentage of subjects | 1.6 | 2.4
Statistical Analysis 1: Comparison: Insulin Degludec (IDeg) vs Insulin Glargine (IGlar); Stepwise hierarchical testing procedure: Step 3: Proportion of subjects with one or more severe hypoglycaemic episodes in the maintenance period; Test type: Superiority or Other; p = 0.3458, McNemar — Superiority was confirmed if the p-value was less than 0.025

4. Secondary Outcome: Incidence of Treatment Emergent Adverse Events
Description: Treatment emergent adverse event was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Time Frame: During 32 weeks of treatment for each treatment period
Population: Safety analysis set included all subjects receiving at least one dose of the investigational product or its comparator (Total number of subjects analysed for this endpoint: 713).
Measure: Number; unit: events
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 671 | 665
events | 1293 | 1381

5. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c (glycosylated haemoglobin) at week 32 (treatment period 1) and at week 64 (treatment period 2). Week 32 HbA1c value was considered as baseline for calculating change from baseline in HbA1c at week 64.
Time Frame: Week 32, Week 64
Population: Full analysis set. Here, 'n' specifies the number of subjects with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg)
Number analyzed (Participants) | 360 | 360
percentage of glycosylated haemoglobin
  week 32 (n=308, 313) | -0.49 (0.99) | -0.58 (1.02)
  week 64 (n=295, 301) | 0.03 (0.75) | 0.10 (0.83)
Statistical Analysis 1: Comparison: Insulin Degludec/Insulin Glargine (IDeg/IGlar) vs Insulin Glargine/Insulin Degludec (IGlar/IDeg); Change from baseline in HbA1c at week 32 (treatment period 1). Before the primary endpoint was tested, the secondary supportive efficacy endpoint "Change from baseline in HbA1c after 32 weeks of treatment" was tested for non-inferiority as prerequisite for testing the primary endpoint. Analysis was performed using a mixed model for repeated measurement (MMRM) with treatment, sex, antidiabetic therapy at screening, visit and dosing time as fixed effects, and age and baseline HbA1c as covariates; Test type: Non-Inferiority or Equivalence — Non-inferiority of IDeg against IGlar was considered confirmed if the upper bound of the two-sided 95% confidence interval was below or equal to 0.40%; Treatment contrast = 0.09, 95% CI 2-sided [-0.04 to 0.23]
Statistical Analysis 2: Comparison: Insulin Degludec/Insulin Glargine (IDeg/IGlar) vs Insulin Glargine/Insulin Degludec (IGlar/IDeg); Change from baseline in HbA1c at week 64 (treatment period 2). The baseline values are week 32 values. Before the primary endpoint was tested, the secondary supportive efficacy endpoint "Change from baseline in HbA1c after 32 weeks of treatment" was tested for non-inferiority as prerequisite for testing the primary endpoint. Analysis was performed using a MMRM with treatment, sex, antidiabetic therapy at screening, visit and dosing time as fixed effects, and age and baseline HbA1c as covariates; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval was below or equal to 0.40%; Treatment contrast = 0.06, 95% CI 2-sided [-0.07 to 0.18]

6. Secondary Outcome: FPG (Fasting Plasma Glucose)
Description: Fasting plasma glucose values at week 32 and week 64.
Time Frame: week 32, week 64
Population: Full analysis set. Here, 'n' specifies the number of subjects with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Degludec/Insulin Glargine (IDeg/IGlar) | Insulin Glargine/Insulin Degludec (IGlar/IDeg)
Number analyzed (Participants) | 360 | 360
mg/dL
  week 32 (n=307, 311) | 107.33 (41.72) | 106.96 (39.81)
  week 64 (n=293, 302) | 114.07 (51.91) | 107.55 (51.30)

ADVERSE EVENTS:
Time Frame: From the first day of exposure to randomised treatment and no later than the last day of randomised treatment (64 weeks)
Description: Subjects in the safety analysis set contributed to the evaluation of adverse events. Treatment emergent adverse event was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Arm/Group | Insulin Degludec (IDeg) | Insulin Glargine (IGlar)
Serious Adverse Events (participants affected / at risk) | 64/671 | 65/665
Other Adverse Events (participants affected / at risk) | 93/671 | 77/665
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec (IDeg) (N=671) | Insulin Glargine (IGlar) (N=665)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 4 (4)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Carpal tunnel decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0)
Confusion postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (9)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lead dislodgement (General disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mitral valve repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 3 (3)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertebral artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec (IDeg) (N=671) | Insulin Glargine (IGlar) (N=665)
Nasopharyngitis (Infections and infestations) | 50 (59) | 41 (49)
Upper respiratory tract infection (Infections and infestations) | 44 (53) | 37 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.